CLINICAL TRIAL: NCT04042376
Title: A Single Arm, Multicenter, Phase 4 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib (PCI-32765) in Chinese Subjects With Relapse or Refractory Waldenström's Macroglobulinemia
Brief Title: A Study of Ibrutinib (PCI-32765) in Chinese Participants With Relapse or Refractory Waldenstrom's Macroglobulinemia (WM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108654; 54179060WAL4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib 420 milligram (mg) (Experimental): Participants will receive ibrutinib 420 mg once daily, continuously starting at Day 1 of Week 1 until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be administered orally, once daily, at a dose of 420 mg (140 mg*3 capsules taken together at one time).
  Other Names: JNJ-54179060; PCI-32765

SUMMARY:
The purpose of this study is to evaluate the efficacy of ibrutinib based on overall response rate (ORR) (partial response [PR] or better) by investigator assessment per the modified Consensus Response Criteria from the Sixth International Workshop on Waldenstrom's Macroglobulinemia (IWWM) (NCCN 2019), in Chinese participants with relapsed or refractory waldenstrom's macroglobulinemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than or equal to (>=) 18 years of age
* Eastern Cooperative Oncology Group (ECOG) less than or equal to (<=) 2
* Previously received at least one prior therapy for WM and have had either documented disease progression or had no response to the most recent treatment regimen
* Centrally confirmed clinicopathological diagnosis of WM
* Measurable disease defined as serum monoclonal immunoglobulin M (IgM) >0.5 gram per deciliter (g/dL)
* Symptomatic disease, requiring treatment
* Hematology and biochemical values within protocol-defined limits
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective methods of contraception while taking study drug. Female participants of childbearing potential should avoid becoming pregnant while taking ibrutinib and for up to 1 month after the last dose of study drug. Male participants must use an effective barrier method of contraception during the study and for 3 months following the last dose of ibrutinib if sexually active with a female of childbearing potential

Exclusion Criteria:

* Involvement of the central nervous system by WM
* Evidence of disease transformation
* Prior exposure to BTK inhibitors
* Known hypersensitivity reaction to ibrutinib or to the excipients in its formulation
* Received any WM-related therapy <=30 days prior to first administration of study treatment
* Received a prior allogeneic hematopoietic stem cell transplant
* Plasmapheresis <35 days prior to the initiation of study drug, except when at least one serum IgM central assessment was performed during the screening period and was >35 days from the most recent plasmapheresis procedure
* History of other malignancies, except: (a) malignancy treated with curative intent and with no known active disease present for >=2 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician; (b) adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease; (c) adequately treated carcinoma in situ without evidence of disease
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Infection requiring systemic treatment that was completed <=14 days before the first dose of study drug
* Bleeding disorders or hemophilia
* Stroke or intracranial hemorrhage within 6 months prior to enrollment
* Infection with human immunodeficiency virus (HIV) or active infection with hepatitis B or hepatitis C
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the participant's safety or put the study outcomes at undue risk
* Currently active, clinically significant hepatic impairment Child-Pugh Class B or C according to the Child Pugh classification
* Currently active, clinically significant cardiovascular disease
* Requires or receiving anticoagulation with warfarin or other Vitamin K antagonists
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
* Lactating or pregnant
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local participant privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- China (6):
  - The First Hospital of Jilin University, Changchun
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Yi S, Cai Z, Hu Y, He A, Gao S, Li Q, Sha L, Zhang N, Ren Y, Gai X, Yang X, Qin R, Qiu L. Ibrutinib Efficacy, Safety, and Pharmacokinetics in Chinese Patients with Relapsed or Refractory Waldenstrom's Macroglobulinemia: A Multicenter, Single-Arm, Phase 4 Study. Adv Ther. 2024 Feb;41(2):672-685. doi: 10.1007/s12325-023-02720-w. Epub 2023 Dec 11. PMID 38079089

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib 420 mg: Participants with relapsed or refractory waldenstrom's macroglobulinemia received ibrutinib 420 milligrams (mg) (3*140 mg capsules) orally once daily from Day 1 of Week 1 until disease progression, unacceptable toxicity, whichever occurs first.
Period: Overall Study
Arm/Group | Ibrutinib 420 mg
Started | 17
Completed | 13
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Not Hispanic or Latino | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved partial response (PR) or better (VGPR) per the modified consensus response criteria from sixth International Workshop on Waldenstrom's Macroglobulinemia (IWWM) (National Comprehensive Cancer Network [NCCN], 2019). PR: greater than or equal to (>=) 50 percent (%) reduction of serum immunoglobulin M (IgM) from baseline, with reduction in lymphadenopathy/splenomegaly if present at baseline. Very Good Partial Response (VGPR): >=90% reduction of serum IgM from baseline or normal serum IgM values, with reduction in lymphadenopathy/splenomegaly if present at baseline.
Time Frame: From start of the treatment (Day 1) up to 49.3 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Percentage of Participants | 70.6 [47.8 to 87.6]

2. Secondary Outcome: Clinical Response Rate (CRR)
Description: CRR was defined as the percentage of participants who achieved minor response (MR) or better according to the modified sixth IWWM (NCCN 2019) criteria as assessed by the investigator. MR: >=25% but less than (<) 50% reduction of serum IgM from baseline.
Time Frame: From start of the treatment (Day 1) up to 49.3 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Percentage of Participants | 100.0 [83.8 to 100.0]

3. Secondary Outcome: Very Good Partial Response (VGPR) or Better Response Rate
Description: VGPR or better response rate was defined as the percentage of participants who achieved VGPR or better according to the modified sixth IWWM (NCCN 2019) criteria as assessed by the investigator. VGPR: >=90% reduction of serum IgM from baseline or normal serum IgM values, with reduction in lymphadenopathy/splenomegaly if present at baseline.
Time Frame: From start of the treatment (Day 1) up to 49.3 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Percentage of Participants | 5.9 [0.3 to 25.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR: duration from date of initial documentation of response (PR/better) to date of first documented progressive disease(PD), death or date of censoring if applicable, for responders (PR/better), as assessed by investigator. VGPR/PR: >=90% reduction or normal serum IgM values (for VGPR) and >=50% (for PR) reduction of serum IgM, with reduction in lymphadenopathy/splenomegaly if present at baseline. PD(at least 1): >=25% IgM increase in serum IgM with >=500 milligrams per deciliters(mg/dL) increase from nadir(lowest serum IgM value at any time from baseline), confirmation needed if IgM was sole PD criterion; new lymph nodes >1.5 centimeters(cm), >=50% increase in nadir in sum of product of diameters; 50% increase in longest diameter of previously identified node >1cm in short axis; new splenomegaly; new extranodal disease; new/recurrent bone marrow involvement; new symptomatic disease(pleural effusion/Bing Neel syndrome/amyloidosis/light chain deposition/paraprotein mediated disorder).
Time Frame: From the date of first documented response up to date of first documented PD or death (Day 1 up to 49.3 months)
Population: Analysis population included responders in all treated analysis set who achieved PR or better.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 12
Months | 20.27 [11.07 to NA] — Here, 'NA' signifies that upper limit of 95% confidence interval could not be estimated due to less number of participants with event.

5. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from the date of first dose to the date of initial documentation of a response (PR or better) for responders. PR: >=50% reduction of serum IgM from baseline, with reduction in lymphadenopathy/splenomegaly if present at baseline. VGPR: >=90% reduction of serum IgM from baseline or normal serum IgM values, with reduction in lymphadenopathy/splenomegaly if present at baseline.
Time Frame: From start of the treatment up to first documentation of PR or better (Day 1 up to 49.3 months)
Population: Analysis population included responders in all treated analysis set who achieved PR or better.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 12
Months | 3.71 [1.84 to 3.71]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as duration from the date of first dose to the date of disease progression or death, whichever occurs first, assessed according to the modified sixth IWWM (NCCN 2019) criteria. PD (at least 1 of the following): >=25% IgM increase in serum IgM with >=500 mg/dL increase from nadir (lowest serum IgM value at any time from baseline), confirmation needed if IgM was sole PD criterion; new lymph nodes >1.5 cm, >=50% increase in nadir in sum of product of diameters; 50% increase in longest diameter of previously identified node >1 cm in short axis; new splenomegaly; new extranodal disease; new/recurrent bone marrow involvement; new symptomatic disease (pleural effusion, Bing Neel syndrome, amyloidosis, light chain deposition, paraprotein mediated disorder).
Time Frame: From day of first dose (Day 1) until PD or death (up to 49.3 months)
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug. Here, 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 9
Months | 23.95 [14.69 to NA] — Here, 'NA' signifies that upper limit of 95% confidence interval could not be estimated due to less number of participants with event.

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was measured from the date of first dose to the date of the participant's death from any cause.
Time Frame: From day of first dose (Day 1) until death due to any cause (up to 49.3 months)
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Months | NA [NA to NA] — Here, 'NA' signifies that median, lower and upper limit of 95% confidence interval could not be estimated due to less number of participants with event.

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Grade 3 or Higher TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were defined as AEs occurring after the first dose of study drugs and within 30 days following the last dose of study drug or initiation of subsequent antineoplastic treatment, whichever occurred earlier. TEAEs were graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03 as Grade 1= Mild; Grade 2= Moderate; Grade 3= Severe; Grade 4= Life-threatening and Grade 5= Death. Number of participants with TEAEs and Grade 3 or higher TEAEs (included serious and non-serious events) were reported in this outcome measure.
Time Frame: From start of the treatment (Day 1) up to 30 days after last dose or initiation of subsequent antineoplastic treatment, whichever occurred first (Day 1 up to 45.9 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Participants
  TEAEs | 17
  Grade 3 or Higher TEAEs | 15

9. Secondary Outcome: Plasma Concentration of Ibrutinib
Description: Plasma concentrations of ibrutinib were reported.
Time Frame: Pre-dose on Day 1 of Weeks 1, 5 and 9
Population: Pharmacokinetics (PK) evaluable analysis set included all enrolled participants who received at least 1 dose of ibrutinib and had at least 1 available PK sample after treatment. Here, 'n' (number analyzed) signifies number of participants evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 17
Nanograms per milliliter (ng/mL)
  Predose Day 1 Week 1: number analyzed (Participants) | 16
  Predose Day 1 Week 1 | NA (NA) — Here, 'NA' signifies that mean and standard deviation could not be calculated as concentration was below quantification limit (<0.500 ng/mL).
  Predose Day 1 Week 5: number analyzed (Participants) | 16
  Predose Day 1 Week 5 | 3.46 (3.97)
  Predose Day 1 Week 9 | 6.27 (8.36)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From Day 1 up to 49.3 months; Serious and other adverse events: From first dose of study drug (Day 1) up to 30 days after last dose of study drug (up to 45.9 months)
Description: All-cause mortality: All treated analysis set included all enrolled participants who received at least 1 dose of study drug. Serious and other adverse events: Safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Ibrutinib 420 mg
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib 420 mg (N=17)
Anal Abscess (Infections and infestations) | 1
Bacterial Prostatitis (Infections and infestations) | 1
Covid-19 Pneumonia (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Lung Squamous Cell Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage Intracranial (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib 420 mg (N=17)
Anaemia (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Ventricular Arrhythmia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Retinal Haemorrhage (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1
Mouth Ulceration (Gastrointestinal disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Anal Abscess (Infections and infestations) | 1
Bacterial Prostatitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 2
Eye Infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes Simplex (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 2
Orchitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 5
Urinary Tract Infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Blood Urea Increased (Investigations) | 1
Hepatitis B DNA Assay Positive (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 5
Platelet Count Decreased (Investigations) | 3
Weight Decreased (Investigations) | 1
Weight Increased (Investigations) | 3
White Blood Cell Count Decreased (Investigations) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage Intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 4
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Scalp Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will delay to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT04042376/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT04042376/SAP_001.pdf